CLINICAL TRIAL: NCT05202054
Title: The Effect of Mindfulness Stress Reduction Program Applied to Postmenopausal Women on Insomnia and Quality of Life
Brief Title: Insomnia and Mindfulness Stress Reduction Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NURDİLAN SENER (Other)
Responsible Party: Sponsor-Investigator, NURDİLAN SENER, principal investigator, Firat University
Organization: Firat University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: FIRAT UNIVERSTY
Record Dates: First submitted 2021-11-22; First posted 2022-01-21 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Postmenopausal Symptoms
Keywords: Menopause; Sleep; QUALITY OF LIFE; NURSING

STUDY DESIGN:
Intervention Model Description: PRETEST POSTTEST EXPERIMENTAL RANDOMIZED STUDY
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of mindfulness stress reduction program on slepness and quality of life (Experimental): Groups of 20 will be formed for the implementation of the mindfulness stress reduction program in the experimental group. The BFSAP day and time will be determined by taking into account the time zones where women are available. 150 minutes of BFSAP will be applied to the women in the experimental group once a week, lasting 8 weeks and consisting of 8 times in total. The women will then be given a midterm test. After the midterm, women will be asked to individually repeat the BFSAP application in their own home for 8 weeks (weeks 8-16).
  Interventions: Other: mindfulness stress reduction program
- control group (No Intervention): THESE PARTICIPANTS HAVE NOT BEEN APPLIED

INTERVENTIONS:
Other: mindfulness stress reduction program — Before the program is implemented, in case women forget, they will be called and reminded of the training time, and they will be invited to the program. The women in the experimental group will be administered 150 minutes of BFSAP once a week, lasting 8 weeks, and consisting of 8 times in total. Afterwards, the women will be given an intermediate test. After the midterm test, women will be asked to individually repeat their BFSAP administration in their own home for 8 weeks (weeks 8-16).
  Arms: The Effect of mindfulness stress reduction program on slepness and quality of life

SUMMARY:
Menopause is the longest life stage in a woman's life, in which psychological and social changes are experienced as well as physical changes and some health problems occur. The symptoms of menopause develop due to varying degrees of somatic and psychological changes that occur as a result of the gradual loss of function of the ovaries. One of the most common and disturbing symptoms of menopause is sleep problems. Sleep is seen as an important health variable that affects an individual's quality of life and well-being. The need for sleep is included among the basic care problems by nursing theorists, and sleep-related problems are included as a nursing diagnosis in the nursing literature. In the literature, it has been stated that mindfulness stress reduction program reduces menopausal symptoms.

Nurses should have knowledge about menopause and coping methods in the field. Although the number of studies examining the effect of mindfulness stress reduction program on insomnia, which is one of the menopausal complaints, is very few in the literature.

DETAILED DESCRIPTION:
Menopause is a medical term defined as the absence of menstrual bleeding lasting more than one year in women in a certain period of life. Menopause is the longest life stage in a woman's life, in which psychological and social changes are experienced as well as physical changes and some health problems occur. The symptoms of menopause develop due to varying degrees of somatic and psychological changes that occur as a result of the gradual loss of function of the ovaries. One of the most common and disturbing symptoms of menopause is sleep problems.

Sleep is accepted as one of the basic physiological needs of humans, which covers 1/3 of human life and ensures the continuity of health. In addition to productivity and efficiency, sleep positively affects cognitive functions such as memory and concentration and contributes to physical and psychological restoration. Because of these positive effects, sleep is seen as an important health variable that affects an individual's quality of life and well-being.

The need for sleep is included among the basic care problems by nursing theorists, and sleep-related problems are included as a nursing diagnosis in the nursing literature. "Discomfort in sleep pattern", which is defined as a condition that causes discomfort in the quality and quantity of the resting pattern or affects the lifestyle, is an important nursing diagnosis that also affects the quality of life and is among the nursing diagnoses determined by NANDA (North American Nursing Diagnosis Association).

In order to cope with the problems participan experience in the menopausal period, women seek various pharmacological and non-pharmacological ways. When the studies conducted in recent years are examined, it has been determined that the commonly used complementary alternative therapies reduce the complaints experienced in menopause. One of the complementary alternative therapies is mindfulness. In the literature, it has been stated that mindfulness stress reduction program reduces menopausal symptoms.

Nurses should have knowledge about menopause and coping methods in the field. Counseling the individual and the family is among the responsibilities of the nurse. Although the number of studies examining the effect of mindfulness stress reduction program and acupuncture on insomnia, which is one of the menopausal complaints, is very few in the literature. It is thought that this study, which was designed to examine the effect of mindfulness stress reduction program on insomnia and quality of life from menopausal complaints, will provide evidence and bring innovation to nursing profession practices.

ELIGIBILITY:
Inclusion Criteria:

* being able to read and write,
* Not having a period for at least a year,
* Not having any diagnosed psychiatric disease or not using medication,
* Not using or not using hormone replacement therapy.

Exclusion Criteria:

* To have entered menopause with surgical methods,
* Not participating in at least two group programs.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only the menopausal period
Enrollment: 192 (Actual)
Dates: Start 2022-04-03 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
women's health initiative insomnia scale | UP TO 16 WEEKS
  Levine et al. (2003) the validity and reliability study of the scale in our country was done by Timur and Şahin (2009). The scale is a Likert type scale consisting of 5 questions. In the study of Timur and Şahin (2009), the Cronbach Alpha value was found to be 0.85.

SECONDARY OUTCOMES:
Menopause-Specific Quality of Life Scale | up to 16 weeks
  The scale was developed by Hilditch et al. in 1996 to measure menopause-specific quality of life. It was adapted to Turkish society by Kharbouch and Şahin in 2005 and its validity and reliability were determined. The scale is a 7-point Likert type scale consisting of 29 questions.
  Each sub-domain score was scored from 0 to 6 in the MCQC. "0" points that there is no problem with that issue. A score of "1" indicates that the problem exists, but this problem is not disturbing at all, while scores between 2-6 indicate the severity and increasing levels of the existing problem. The lowest score that can be obtained from the scale is 0, the highest score is 174. The scale consists of four sub-dimensions: vasomotor, psychosocial, physical and sexual. As the score increases, the severity of the complaint increases and the quality of life decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- NURDİLAN, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sener Cetin N, Nacar G, Timur Tashan S. The effect of mindfulness-based stress reduction program applied to postmenopausal women on insomnia and quality of life. Women Health. 2024 Aug;64(7):573-583. doi: 10.1080/03630242.2024.2382420. Epub 2024 Jul 28. PMID 39069644